CLINICAL TRIAL: NCT04785131
Title: The Impact of Consuming California Dried Plums on Bone Health of Young Women Using Hormonal Contraceptives
Brief Title: Prune Consumption and Bone Health in Young Women Using Hormonal Contraceptives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Shirin Hooshmand, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 59871A
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Osteoporosis Risk
Keywords: Prune; Bone health; Oral contraceptives; Women health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prune group (Experimental): Oral contraceptive users will consume 50 grams prunes daily.
  Interventions: Other: Prune
- Oral contraceptive users (No Intervention): Oral contraceptive users will be monitored throughout the study period.
- Non oral contraceptive users (No Intervention): Non oral contraceptive users will be monitored throughout the study period.

INTERVENTIONS:
Other: Prune — daily consumption of 50 grams prune.
  Arms: Prune group

SUMMARY:
The primary objective of this study is to determine if 12 months of consuming 50 grams of dried plum daily will prevent bone loss or augment bone accrual of young adult oral contraceptive (OC) users.

DETAILED DESCRIPTION:
Eligible participants will be assigned among three groups 1) control non-OC users, 2) control OC users, and 3) dried plum OC users. OC users will be randomly allocated to the dried plum OC group, which will consume 50 g dried plum daily for 12 months, or a control group, for which dried plums will not be allowed and no control food will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25

Exclusion Criteria:

* Metabolic bone disease, renal disease, cancer, CVD, diabetes mellitus, respiratory disease, gastrointestinal disease, liver disease or other chronic diseases, heavy smoking (more than twenty cigarettes/day) and current use of any prescription medications known to alter bone and calcium metabolism
* Regularly consumed dried plum or prune juice

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in bone mineral density from baseline to 12 months | At baseline, at 12 months
  Bone density measurements with DXA

SECONDARY OUTCOMES:
Changes from baseline in bone specific alkaline phosphatase at 6 months and 12 months | At baseline, at 6 months, at 12 months
  Bone biomarkers measurements with ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Hooshmand, PhD, RD, Study Director — San Diego State University
Locations (2):
- United States (2):
  - Shirin Hooshmand, San Diego, California
  - School of Exercise and Nutritional Sciences, San Diego, California

REFERENCES:
- [Derived] DeMasi T, Tsang M, Mueller J, Giltvedt K, Nguyen TN, Kern M, Hooshmand S. Prunes May Blunt Adverse Effects of Oral Contraceptives on Bone Health in Young Adult Women: A Randomized Clinical Trial. Curr Dev Nutr. 2024 Jul 18;8(9):104417. doi: 10.1016/j.cdnut.2024.104417. eCollection 2024 Sep. PMID 39310666